CLINICAL TRIAL: NCT01146145
Title: Efficacity, Safety and Cost of Intravenous Morphine Titration Alone or Combined to Ketamine
Acronym: KEMO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Zakia IDIR, Department Clinical Research of Developpemnt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P020401
Record Dates: First submitted 2010-06-16; First posted 2010-06-17 (Estimated); Last update posted 2010-06-17 (Estimated); Status verified 2010-06

CONDITIONS: Postoperative Pain
Keywords: postoperative; pain; analgesia; morphine; titration; ketamine
MeSH Terms: conditions — Pain, Postoperative; Pain; Agnosia | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- treatment (Experimental): intravenous morphine titration combined to ketamine
  Interventions: Drug: Ketamine
- placebo (Placebo Comparator): morphine titration alone
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — intravenous morphine titration combined to ketamine
  Other Names: two groups of patients recevieving; in the postanesthesia care unit either; intravenous morphine titration alone; or intravenous morphine titration combined to ketamine

SUMMARY:
This is a randomised, controlled, double blinded study comparing in the postoperative setting the analgesic efficacy, the safety and the cost in two groups of patients receiving in the postanesthesia care unit either intravenous morphine titration alone or intravenous morphine titration combined to ketamine.

DETAILED DESCRIPTION:
Randomised, controlled, double blinded study comparing in the postoperative setting the analgesic efficacy, the safety and the cost in two groups of patients receiving in the postanesthesia care unit either intravenous morphine titration alone or intravenous morphine titration combined to ketamine

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 yrs
* scheduled surgery
* General anesthesia
* ASA I to III
* Able to use a VAS
* No psychological disorders, able to speak french

Exclusion Criteria:

* Age < 18 yrs
* Locoregional anesthesia or analgesia
* Allergia to morphine or ketamine
* Morphine or ketamine contraindication
* Pregnancy or breast-feeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2003-05; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
analgesic efficacy | 24 h
  the analgesic efficacy, in two groups of patients recevieving in the postanesthesia care unit either intravenous morphine titration alone or intravenous morphine titration combined to ketamine

CONTACTS AND LOCATIONS:
Overall Officials: Hawa Keita, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hopital Louis Mourier, Colombes, France